CLINICAL TRIAL: NCT06158334
Title: Study of Surgical Practices in Patient With Haemophilia A or B Treated With an Extended Half-life Recombinant Factor VIII-Fc or IX-Fc (ELOCTA®, ALPROLIX®)
Brief Title: Study of Surgical Practices in Patients With Haemophilia A or B Treated With an Extended Half-life Recombinant Factor VIII-Fc or IX-Fc (ELOCTA®, ALPROLIX®)
Acronym: CHALE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 868
Record Dates: First submitted 2023-06-19; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: surgery; Haemophilia A; Haemophilia B; Elocta®; Alprolix®
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Minor and major surgeries of patients with haemophilia A treated with Elocta®: Description of all surgical data (minor and major) on Elocta® (all dosage and treatment regimens)
  Interventions: Drug: Describe the respective haemostatic efficacy of Elocta® for haemopilia A during surgical procedures
- Minor and major surgeries of patients with haemophilia B treated with Alprolix®: Description of all surgical data (minor and major) on Alprolix® (all dosage and treatment regimens)
  Interventions: Drug: Describe the respective haemostatic efficacy of Alprolix® for haemopilia B during surgical procedures

INTERVENTIONS:
Drug: Describe the respective haemostatic efficacy of Elocta® for haemopilia A during surgical procedures — All surgical data will be collected: surgery, biology, administration of Elocta®, bleeding and transfusion, hemostatic efficacity, surgery complication and bleeding
  Groups: Minor and major surgeries of patients with haemophilia A treated with Elocta®
Drug: Describe the respective haemostatic efficacy of Alprolix® for haemopilia B during surgical procedures — All surgical data will be collected: surgery, biology, administration of Alprolix®, bleeding and transfusion, hemostatic efficacity, surgery complication and bleeding…
  Groups: Minor and major surgeries of patients with haemophilia B treated with Alprolix®

SUMMARY:
Haemophilia A and haemophilia B are inherited bleeding disorders resulting from the absence or deficiency of coagulation factors VIII and IX, respectively. The peri-operative period of people with haemophilia is commonly managed with replacement therapy.

In phase 3 studies of Elocta® (extended half-life recombinant factor VIII-Fc) and Alprolix® (extended half-life recombinant factor IX-Fc), haemostatic efficacy was demonstrated to be good or excellent, close to the haemostatic efficacy usually seen in people without haemophilia, with maintenance and stability of circulating FVIII and FIX levels compatible with the surgical procedure, while reducing the frequency of infusions and consumption of therapeutic units. In 2019, the National Protocol for Diagnosis and Care in haemophilia recommended 2 methods for managing patients with haemophilia in the peri-operative period, either discontinuous injections of standard or extended half-life factor VIII/IX or a continuous infusion of FVIII/IX.

Many countries, including France, have adopted these rFVIII/IXFc therapeuitic products and recommended their use in the surgical management of patients. However, the use of these two products in real life during surgery in haemophilic A and B patients has not been described in detail. It seems therefore relevant to better document their use in order to progressively specify their use during surgeries with varied bleeding risks.

ELIGIBILITY:
Inclusion Criteria:

* patient with Haemophilia A or B
* surgery performed with Elocta® or Alprolix®
* Information leaflet given to the patient who as reached the age of majority or to the parents or legal guardian for minors

Exclusion Criteria:

* Any blood coagulation disorder other than Haemophilia A or B
* Patient with factor VIII or IX inhibitor
* Severe liver disease (serum ALAT/ASAT levels> 5 x ULN)
* Severe renal disease (serum creatinine > 2x ULN)
* Known hypersensitivity to the substances or its excipients
* patient participating in another clinical trial or having participated in another clinical trial within the previous 30 days (non-interventional studies are not a criterion for non-inclusion)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (minor and adults) with Haemophilia A or B for whom minor and major surgeries is performed with Elocta® or Alprolix®.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative haemostatic efficacy described in real life with ELOCTA® and ALPROLIX® in haemophilia A and B patients. Haemostatic efficacy is defined by excellent, good, fair, poor. | 15 days post-surgery
  changes in hemostatic efficacy between surgery and 15 days post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence en Hémophilie, hôpityal Louis Pradel, GHE- Hospices Civils de Lyon, Bron, France